CLINICAL TRIAL: NCT06035393
Title: A Phase II, Randomized, Double Blind, Double Dummy, Active-controlled, Parallel-group Study to Assess the Efficacy and Safety of HRG2005 Inhalation in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Assess the Efficacy and Safety of HRG2005 Inhalation in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's R&D strategy adjusted.
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRG2005-201
Record Dates: First submitted 2023-09-07; First posted 2023-09-13 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Intervention Model Description: This is a randomized, double blind, double dummy, active-controlled, parallel-group study.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A (Experimental): Drug1 dose 1+Drug 3
  Interventions: Drug: HRG2005 inhalation; Drug: Placebo to match Indacaterol Maleate and Glycopyrronium Bromide Powder for inhalation
- Treatment group B (Experimental): Drug1 dose 2+Drug 2+Drug 3
  Interventions: Drug: HRG2005 inhalation; Drug: Placebo to match HRG2005 inhalation; Drug: Placebo to match Indacaterol Maleate and Glycopyrronium Bromide Powder for inhalation
- Treatment group C (Experimental): Drug1 dose 3+Drug 2+Drug 3
  Interventions: Drug: HRG2005 inhalation; Drug: Placebo to match HRG2005 inhalation; Drug: Placebo to match Indacaterol Maleate and Glycopyrronium Bromide Powder for inhalation
- Treatment group D (Other): Drug 2+Drug 4
  Interventions: Drug: Placebo to match HRG2005 inhalation; Drug: Indacaterol Maleate and Glycopyrronium Bromide Powder for inhalation

INTERVENTIONS:
Drug: HRG2005 inhalation — Drug 1: dose 1; dose 2; dose 3
  Arms: Treatment group A; Treatment group B; Treatment group C
Drug: Placebo to match HRG2005 inhalation — Drug 2
  Arms: Treatment group B; Treatment group C; Treatment group D
Drug: Placebo to match Indacaterol Maleate and Glycopyrronium Bromide Powder for inhalation — Drug 3
  Arms: Treatment group A; Treatment group B; Treatment group C
Drug: Indacaterol Maleate and Glycopyrronium Bromide Powder for inhalation — Drug 4
  Arms: Treatment group D

SUMMARY:
This is a randomized, double blind, double dummy, active-controlled, parallel-group study to assess the efficacy and Safety of HRG2005 inhalation in patients with moderate to severe chronic obstructive pulmonary disease. Approximately 200 patients with moderate to severe COPD will be randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the study protocol;
2. Subjects 40 years of age or older (inclusive), Male or female subjects;
3. Subjects with an established clinical history of COPD;
4. A post-bronchodilator FEV1/FVC ratio must be <0.7 at Screening and FEV1 must be <80% and ≥30% predicted normal at pre-randomization;
5. a documented history of ≥ 2 moderate or ≥ 1 severe COPD exacerbation in the previous 12 months;
6. Tobacco Use: Current or former smokers with a history of at least 10 pack-years of cigarette smoking;
7. A score of ≥10 on the COPD Assessment Test (CAT) at pre-randomization.

Exclusion Criteria:

1. Subjects who required systemic corticosteroids or antibiotics or hospitalized due to poorly controlled COPD or who had lower respiratory tract infections that required antibiotics within 4 weeks prior to Screening to pre-randomization;
2. Subjects who had respiratory tract infections that required antibiotics within 2 weeks prior to Screening to pre-randomization;
3. Subjects with other respiratory or respiratory related diseases, including but not limited to asthma, active tuberculosis, lung cancer, interstitial pulmonary disease, α1-antitrypsin deficiency, pulmonary heart disease, clinically significant pulmonary hypertension, clinically significant bronchiectasis, or other active pulmonary disease;
4. Subjects with lung volume reduction surgery within the 12 months prior to Screening;
5. Subjects who have Other known serious medical conditions；
6. Subjects receiving oxygen therapy required for greater than 15 hours a day;
7. Clinically significant electrocardiogram abnormality；
8. Subjects with significant laboratory abnormality at screening；
9. Suspected allergy to any ingredient in the study drug;
10. Participation in clinical trials of any drug or medical device (except for screening failures) within 4 weeks before screening, or within 5 half-lives of the drug at screening (whichever is longer);
11. Pregnant or lactating females;
12. History of drug abuse within one year before screening
13. Other conditions judged by the investigator to be not suitable to participate in the trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in morning pre-dose trough FEV1 at week 12 | Up to week 12

SECONDARY OUTCOMES:
Change from baseline in morning pre-dose trough FEV1 at each time point | up to week 48
Compared with the active-controlled group in morning pre-dose trough FEV1 at each time point | up to week 48
Proportion of subjects achieving an improvement from baseline≥100mL in morning pre-dose trough FEV1 | up to week 48
Peak change from baseline in FEV1 at week 12 | Up to week 12
FEV1 area under the curve from 0 to 12 hours (AUC0-12), 0 to 24 (AUC0-24) hours at Week 12 | Up to week 12
Rate of moderate or severe COPD exacerbations over 48 Weeks | up to week 48
Rate of severe COPD exacerbations over 48 Weeks | up to week 48
Change from baseline in CAT (COPD Assessment test) total score at each time point | up to week 48
Percentage of Days with No Rescue use and change from baseline in average daily rescue use at each time point | up to week 48
Incidence and severity of adverse events | Up to week 50

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided